CLINICAL TRIAL: NCT05447780
Title: Comparing the General Anesthesia, the General Anesthesia With the ESP Block or TLIP Block in the Patients Undergoing Lumbar Surgeries
Brief Title: Comparing General Anesthesia, General Anesthesia With ESP Block or TLIP Block in Patients Undergoing Lumbar Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anesthesia Research Group UA (Other)
Responsible Party: Principal Investigator, Plechysta Yelyzaveta, Chief of the anesthesia department, Anesthesia Research Group UA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1718042022
Record Dates: First submitted 2022-06-17; First posted 2022-07-07 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Disc Herniation; Lumbar Discogenic Pain; Lumbar Spinal Stenosis; Failed Back Surgery Syndrome
MeSH Terms: conditions — Intervertebral Disc Displacement; Spinal Stenosis; Failed Back Surgery Syndrome | interventions — Anesthesia, Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia (Experimental): induction: propofol 1.5-2.5 mg\kg IV bolus and fentanyl 1-2 mcg\kg maintenance anesthesia: sevoflurane, doses of the inhalation agent according to bispectral index (BIS) monitor ( target BIS level 40-60) and fentanyl 1-5 mcg\kg\h.
  Interventions: Procedure: regional anesthesia
- Combined anesthesia: general anesthesia and Erector spinae plane block (ESP block) (Experimental): induction: propofol 1.5-2.5 mg\kg IV bolus and fentanyl 1-2 mcg\kg ESP- block with US control with single shot of local anesthetic ( bupivacaine 0.375% or 0.25% 20-30 ml) is performed after induction.
  maintenance anesthesia: sevoflurane, doses of the inhalation agent according to BIS monitor ( target BIS level 40-60) and fentanyl 0.5-1.5 mcg\kg\h.
  Interventions: Procedure: regional anesthesia
- Combined anesthesia: General anesthesia and Thoraco-lumbar interfacial plane block (TLIP block) (Experimental): induction: propofol 1.5-2.5 mg\kg IV bolus and fentanyl 1-2 mcg\kg TLIP- block with US control with single shot of local anesthetic ( bupivacaine 0.25% 15 ml or mixed bupivacaine 0.25% 7.5 ml and lidocaine 2% 7.5 ml) is performed after induction.
  maintenance anesthesia: sevoflurane, doses of the inhalation agent according to BIS monitor ( target BIS level 40-60) and fentanyl 0.5-1.5 mcg\kg\h.
  Interventions: Procedure: regional anesthesia

INTERVENTIONS:
Procedure: regional anesthesia — regional anesthesia in lumbar surgery, TLIP block in spinal surgery, ESP block in spinal surgery

SUMMARY:
The regional methods of anesthesia for the neurosurgical operations of the spine and spinal cord reducing the needs for opioids intra operatively and reducing pain in the postoperative period, decrease the numbers of failed back syndrome.

ELIGIBILITY:
Inclusion Criteria:

* back surgery

Exclusion Criteria:

* contraindications to the regional method of analgesia,
* patient refusal,
* patients with diabetes mellitus
* mental illness
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
A Visual Analogue Scale (numerical rating scale (NRS) | 2 hours after surgery
  minimum 0 ( no pain), maximum 10 (the worst pain ever)
A Visual Analogue Scale (numerical rating scale (NRS) | 6 hours after surgery
  minimum 0 ( no pain), maximum 10 (the worst pain ever)
A Visual Analogue Scale (numerical rating scale (NRS) | 24 hour after surgery
  minimum 0 ( no pain), maximum 10 (the worst pain ever)
A Visual Analogue Scale (numerical rating scale (NRS) | 48 hour after surgery
  minimum 0 ( no pain), maximum 10 (the worst pain ever)

SECONDARY OUTCOMES:
A Visual Analogue Scale (numerical rating scale (NRS) | 1 month after surgery
  minimum 0 ( no pain), maximum 10 (the worst pain ever)
A Visual Analogue Scale (numerical rating scale (NRS) | 3 month after surgery
  minimum 0 ( no pain), maximum 10 (the worst pain ever)

CONTACTS AND LOCATIONS:
Overall Officials: Yelyzaveta Plechystaya, MD, Study Chair — chief of the anesthesia department
Locations (1):
- Anesthesia department Medical Network Dobrobut, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No